CLINICAL TRIAL: NCT03438708
Title: "PADRES" (Prior Axitinib as a Determinant of Outcome of REnal Surgery)
Brief Title: Prior Axitinib as a Determinant of Outcome of Renal Surgery
Acronym: PADRES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Aditya Bagrodia, Professor of Urology and Radiology, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161197; WI209751 (Other Grant/Funding Number: Pfizer Inc)
Record Dates: First submitted 2018-01-19; First posted 2018-02-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Axitinib; Nephrectomy; Neoadjuvant; Clear Cell Renal Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axitinib Oral Tablet [Inlyta] (Experimental): Axitinib 5 mg PO BID for 8-10 weeks
  Interventions: Drug: Axitinib Oral Tablet [Inlyta]

INTERVENTIONS:
Drug: Axitinib Oral Tablet [Inlyta] — Axitinib 5 milligrams (mg) administered orally (po) twice daily (BID) for 8 weeks (with titration to 7 mg BID as tolerated at 4 weeks)
  Other Names: Inlyta

SUMMARY:
This is a single arm phase II study of axitinib in patients with clear cell renal cell carcinoma (RCC) with strong indications for partial nephrectomy (PN) for whom PN is not currently possible due to anatomic considerations and residual renal function concerns. Evaluation of tumor downsizing will be performed including changes of tumor complexity by nephrometry score. A total of 50 participants will be enrolled.

It is hypothesized that pretreatment with axitinib will be safe and improve the feasibility of complex nephron sparing surgery in select patients with localized clear cell RCC and imperative indications for partial nephrectomy.

DETAILED DESCRIPTION:
The primary objective of the study is to prospectively assess utility of axitinib in facilitation of partial nephrectomy where partial nephrectomy was not thought to be safe/possible in the setting of imperative indication for complex renal masses in renal cell cancer.

Secondary objectives: To determine the safety, tumor diameter (per RECIST v1.1) volume change, surgical morbidity and renal functional outcomes following neoadjuvant axitinib for RCC.

Anatomical/morphometric:

1. tumor diameter/volume change,
2. conversion of hilar to non-hilar tumors,
3. reduction in RENAL morphometric score.

Functional Considerations:

1. Requirement of acute dialysis
2. Change in Glomerular Filtration Rate (GFR)
3. Whether or not GFR crosses 30 threshold, or decline by GFR to >50% of baseline.

Safety indices:

1. Incidence of Clavien >3 complications
2. Avoidance of need for multiple blood transfusions

ELIGIBILITY:
Inclusion Criteria:

1. Localized clear cell renal carcinoma without evidence of distant metastases
2. Imperative indication for nephron sparing surgery

   * Baseline chronic kidney disease (CKD) (stage 3, GFR <60 ml/min/1.73m2), or anatomically or functional solitary kidney (defined by renal scintigraphy of contralateral renal unit with <15% function) or bilateral synchronous disease); and
   * RENAL score ≥10 or proximity to renal hilum (defined as <2 mm away from at least 2 renal hilar vessels-the main artery/vein or first order branches); and
   * Radical nephrectomy would lead to severe CKD (stage 3b, GFR <45 ml/min/1.73m2).
3. Male or female, age ≥ 18 years
4. Karnofsky performance status ≥ 70.
5. Adequate organ function as defined by:

   * Absolute neutrophil count (ANC) ≥1,000/μL
   * Platelets ≥100,000/μL
   * Hemoglobin ≥9.0 g/dL
   * Serum calcium ≤12.0 mg/dL
   * Serum creatinine ≤1.5 x upper limit of normal (ULN)
   * Total serum bilirubin ≤1.5 x ULN
   * SGOT≤2.5 x ULN and serum glutamic pyruvic transaminase (SGPT) ≤2.5x ULN
6. Signed informed consent and willingness/ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

1. Presence of metastatic disease on radiographic imaging.
2. Elective indication for nephron sparing surgery
3. Non-clear cell histology
4. Prior systemic treatment of any kind or radiotherapy for RCC
5. NCI CTCAE Version 5.0 grade 3 hemorrhage within 4 weeks of starting the study treatment
6. Ongoing cardiac dysrhythmias of NCI CTCAE Version 5.0 grade ≥2. Controlled atrial fibrillation is permitted. Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on screening EKG >480 msec.
7. Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal,or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate.
8. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
9. Uncontrolled hypertension (HTN): systolic blood pressure ≥150 or diastolic blood pressure ≥ 100 mmHg or both despite appropriate therapy.
10. HTN with need for greater than three anti-hypertensive agents at baseline. Drug formulations containing two or more anti-hypertensive agents will be counted based on the number of active agents in each formulation.
11. New York Heart Association (NYHA) class III or greater congestive heart failure (CHF)
12. Uncontrolled hyper- or hypothyroidism.
13. Subjects with arterial thrombotic events in the prior 12 months (axitinib has never been studied in this population)
14. Subjects who have had venous thrombotic events in the prior 6 months (axitinib has never been studied in this population)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Percent reduction of longest diameter of tumor in millimeters | 90 days
  Measured by CT or MRI
Objective Tumor Response Rate (by RECIST criteria) | 90 days
  Percentage of patients achieving partial response (reduction in tumor diameter by at least 30% of maximum diameter) as defined by RECIST criteria
Effect on tumor morphometry, as measured by RENAL score [(R)adius, (E)xophytic/endophytic components, (N)earness to the collecting system or sinus, (A)neterior/posterior, and (L)ocation relative to polar lines] | 90 days
  The RENAL nephrometry score quantifies tumor size and location relative to the major blood vessel and collecting system supply of the kidney according to 5 domains (tumor radius, exophytic/endophytic appearance, proximity to urinary collecting system, anterior/posterior location, and location with respect to renal poles). Four of these domains have a score of 1-3, with 3 indicating a more complex score within the domain. The total score is the sum of all of the domains (total minimum score being 4 and the maximum score being 12, and with more complex tumors having a higher score). The study will record effect of the medication on tumor complexity as measured by total RENAL nephrometry score.
Feasibility of partial nephrectomy surgery | 90 days
  Percentage of Successful partial nephrectomy perfomed (as opposed to radical nephrectomy) with negative surgical margins determined by pathological assessment of resection margins.

CONTACTS AND LOCATIONS:
Overall Officials: Ithaar H Derweesh, MD, Study Chair — UC San Diego Moores Cancer Center; Ithaar H Derweesh, MD, Principal Investigator — UC San Diego Moores Cancer Center; Brian I Rini, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center; Steven C Campbell, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rini BI, Campbell SC, Escudier B. Renal cell carcinoma. Lancet. 2009 Mar 28;373(9669):1119-32. doi: 10.1016/S0140-6736(09)60229-4. Epub 2009 Mar 5. PMID 19269025
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] Russo P. End stage and chronic kidney disease: associations with renal cancer. Front Oncol. 2012 Apr 2;2:28. doi: 10.3389/fonc.2012.00028. eCollection 2012. PMID 22649783
- [Background] Kane CJ, Mallin K, Ritchey J, Cooperberg MR, Carroll PR. Renal cell cancer stage migration: analysis of the National Cancer Data Base. Cancer. 2008 Jul 1;113(1):78-83. doi: 10.1002/cncr.23518. PMID 18491376
- [Background] Lee HJ, Liss MA, Derweesh IH. Outcomes of partial nephrectomy for clinical T1b and T2 renal tumors. Curr Opin Urol. 2014 Sep;24(5):448-52. doi: 10.1097/MOU.0000000000000081. PMID 24921904
- [Background] Brandao LF, Zargar H, Autorino R, Akca O, Laydner H, Samarasekera D, Krishnan J, Haber GP, Stein RJ, Kaouk JH. Robot-assisted partial nephrectomy for >/= 7 cm renal masses: a comparative outcome analysis. Urology. 2014 Sep;84(3):602-8. doi: 10.1016/j.urology.2014.04.015. Epub 2014 Jun 12. PMID 24929947
- [Background] Karellas ME, O'Brien MF, Jang TL, Bernstein M, Russo P. Partial nephrectomy for selected renal cortical tumours of >/= 7 cm. BJU Int. 2010 Nov;106(10):1484-7. doi: 10.1111/j.1464-410X.2010.09405.x. PMID 20518765
- [Background] Breau RH, Crispen PL, Jimenez RE, Lohse CM, Blute ML, Leibovich BC. Outcome of stage T2 or greater renal cell cancer treated with partial nephrectomy. J Urol. 2010 Mar;183(3):903-8. doi: 10.1016/j.juro.2009.11.037. Epub 2010 Jan 18. PMID 20083271
- [Background] Long CJ, Canter DJ, Kutikov A, Li T, Simhan J, Smaldone M, Teper E, Viterbo R, Boorjian SA, Chen DY, Greenberg RE, Uzzo RG. Partial nephrectomy for renal masses >/= 7 cm: technical, oncological and functional outcomes. BJU Int. 2012 May;109(10):1450-6. doi: 10.1111/j.1464-410X.2011.10608.x. Epub 2012 Jan 5. PMID 22221502
- [Background] Kopp RP, Mehrazin R, Palazzi KL, Liss MA, Jabaji R, Mirheydar HS, Lee HJ, Patel N, Elkhoury F, Patterson AL, Derweesh IH. Survival outcomes after radical and partial nephrectomy for clinical T2 renal tumours categorised by R.E.N.A.L. nephrometry score. BJU Int. 2014 Nov;114(5):708-18. doi: 10.1111/bju.12580. Epub 2014 Oct 3. PMID 24274650
- [Background] Alanee S, Nutt M, Moore A, Holland B, Dynda D, Wilber A, El-Zawahry A. Partial nephrectomy for T2 renal masses: contemporary trends and oncologic efficacy. Int Urol Nephrol. 2015 Jun;47(6):945-50. doi: 10.1007/s11255-015-0975-3. Epub 2015 Apr 12. PMID 25864101
- [Background] Kopp RP, Liss MA, Mehrazin R, Wang S, Lee HJ, Jabaji R, Mirheydar HS, Gillis K, Patel N, Palazzi KL, Wan JY, Patterson AL, Derweesh IH. Analysis of Renal Functional Outcomes After Radical or Partial Nephrectomy for Renal Masses >/=7 cm Using the RENAL Score. Urology. 2015 Aug;86(2):312-9. doi: 10.1016/j.urology.2015.02.067. Epub 2015 Jul 16. PMID 26189330
- [Background] Randall JM, Millard F, Kurzrock R. Molecular aberrations, targeted therapy, and renal cell carcinoma: current state-of-the-art. Cancer Metastasis Rev. 2014 Dec;33(4):1109-24. doi: 10.1007/s10555-014-9533-1. PMID 25365943
- [Background] Thomas AA, Rini BI, Lane BR, Garcia J, Dreicer R, Klein EA, Novick AC, Campbell SC. Response of the primary tumor to neoadjuvant sunitinib in patients with advanced renal cell carcinoma. J Urol. 2009 Feb;181(2):518-23; discussion 523. doi: 10.1016/j.juro.2008.10.001. Epub 2008 Dec 18. PMID 19100579
- [Background] Cowey CL, Amin C, Pruthi RS, Wallen EM, Nielsen ME, Grigson G, Watkins C, Nance KV, Crane J, Jalkut M, Moore DT, Kim WY, Godley PA, Whang YE, Fielding JR, Rathmell WK. Neoadjuvant clinical trial with sorafenib for patients with stage II or higher renal cell carcinoma. J Clin Oncol. 2010 Mar 20;28(9):1502-7. doi: 10.1200/JCO.2009.24.7759. Epub 2010 Feb 16. PMID 20159822
- [Background] Silberstein JL, Millard F, Mehrazin R, Kopp R, Bazzi W, DiBlasio CJ, Patterson AL, Downs TM, Yunus F, Kane CJ, Derweesh IH. Feasibility and efficacy of neoadjuvant sunitinib before nephron-sparing surgery. BJU Int. 2010 Nov;106(9):1270-6. doi: 10.1111/j.1464-410X.2010.09357.x. PMID 20394613
- [Background] Rini BI, Plimack ER, Takagi T, Elson P, Wood LS, Dreicer R, Gilligan T, Garcia J, Zhang Z, Kaouk J, Krishnamurthi V, Stephenson AJ, Fergany A, Klein EA, Uzzo RG, Chen DY, Campbell SC. A Phase II Study of Pazopanib in Patients with Localized Renal Cell Carcinoma to Optimize Preservation of Renal Parenchyma. J Urol. 2015 Aug;194(2):297-303. doi: 10.1016/j.juro.2015.03.096. Epub 2015 Mar 23. PMID 25813447
- [Background] Karam JA, Devine CE, Urbauer DL, Lozano M, Maity T, Ahrar K, Tamboli P, Tannir NM, Wood CG. Phase 2 trial of neoadjuvant axitinib in patients with locally advanced nonmetastatic clear cell renal cell carcinoma. Eur Urol. 2014 Nov;66(5):874-80. doi: 10.1016/j.eururo.2014.01.035. Epub 2014 Feb 7. PMID 24560330
- [Background] Lane BR, Derweesh IH, Kim HL, O'Malley R, Klink J, Ercole CE, Palazzi KL, Thomas AA, Rini BI, Campbell SC. Presurgical sunitinib reduces tumor size and may facilitate partial nephrectomy in patients with renal cell carcinoma. Urol Oncol. 2015 Mar;33(3):112.e15-21. doi: 10.1016/j.urolonc.2014.11.009. Epub 2014 Dec 19. PMID 25532471
- [Background] Rini BI, Escudier B, Tomczak P, Kaprin A, Szczylik C, Hutson TE, Michaelson MD, Gorbunova VA, Gore ME, Rusakov IG, Negrier S, Ou YC, Castellano D, Lim HY, Uemura H, Tarazi J, Cella D, Chen C, Rosbrook B, Kim S, Motzer RJ. Comparative effectiveness of axitinib versus sorafenib in advanced renal cell carcinoma (AXIS): a randomised phase 3 trial. Lancet. 2011 Dec 3;378(9807):1931-9. doi: 10.1016/S0140-6736(11)61613-9. Epub 2011 Nov 4. PMID 22056247
- [Background] Tzogani K, Skibeli V, Westgaard I, Dalhus M, Thoresen H, Slot KB, Damkier P, Hofland K, Borregaard J, Ersboll J, Salmonson T, Pieters R, Sylvester R, Mickisch G, Bergh J, Pignatti F. The European Medicines Agency approval of axitinib (Inlyta) for the treatment of advanced renal cell carcinoma after failure of prior treatment with sunitinib or a cytokine: summary of the scientific assessment of the committee for medicinal products for human use. Oncologist. 2015 Feb;20(2):196-201. doi: 10.1634/theoncologist.2014-0177. Epub 2015 Jan 23. PMID 25616431
- [Background] Lane BR, Demirjian S, Derweesh IH, Takagi T, Zhang Z, Velet L, Ercole CE, Fergany AF, Campbell SC. Survival and Functional Stability in Chronic Kidney Disease Due to Surgical Removal of Nephrons: Importance of the New Baseline Glomerular Filtration Rate. Eur Urol. 2015 Dec;68(6):996-1003. doi: 10.1016/j.eururo.2015.04.043. Epub 2015 May 23. PMID 26012710
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] van der Veldt AA, Meijerink MR, van den Eertwegh AJ, Bex A, de Gast G, Haanen JB, Boven E. Sunitinib for treatment of advanced renal cell cancer: primary tumor response. Clin Cancer Res. 2008 Apr 15;14(8):2431-6. doi: 10.1158/1078-0432.CCR-07-4089. PMID 18413834